CLINICAL TRIAL: NCT00534651
Title: Paracetamol and Endothelial Function in Patients With Stable Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EK1265
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Coronary Arteriosclerosis; Endothelial Function
MeSH Terms: conditions — Coronary Artery Disease | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Paracetamol — Paracetamol 3x1000mg daily or Placebo for two weeks in a crossover design with a two-week washout-phase in between.

SUMMARY:
The purpose of this study is to determine the effect of orally given paracetamol on the vascular function and on 24-hour blood pressure in patients with coronary artery disease

DETAILED DESCRIPTION:
Patients with chronic pain diseases (e.g. osteoarthritis) are dependent on effective medication. NSAIDs are very effective in lowering pain in these patients. Recently there has aroused major concern with regard to cardiovascular side effects and safety, especially in selective cyclooxygenase-2 inhibitors (coxibs) but also in "regular" NSAIDs.

At the moment, there is a big confusion, whether these drugs still should be used, especially in patients with known coronary artery disease. Physicians now try to switch to high dose paracetamol, despite the weaker efficacy in pain relieve, because this drug is considered generally as not harmful.

As there is very few information on the cardiovascular effect of this drug, we plan to perform this study and investigate the impact of paracetamol on endothelial function, an important cardiovascular surrogate marker, on inflammatory markers and on oxidative stress in patients with coronary artery disease on top of standard medication, including aspirin

ELIGIBILITY:
Inclusion Criteria:

* Age: 30 - 80 years
* History of coronary artery disease (documented by coronary angiogram, nuclear imaging, positive stress test)
* Stable cardiovascular medication for at least 1 month
* Written obtained informed consent

Exclusion Criteria:- myocardial infarction, unstable angina, stroke within 3 months prior to study entry

* coronary intervention/revascularisation procedure within 3 months prior to study entry
* Left ventricular ejection fraction <50%
* Other analgesics (Platelet inhibition therapy with Aspirin 100mg/d will be continued)
* Long acting nitrates
* Smoking
* Chronic heart failure (> NYHA II)
* Ventricular tachyarrhythmias
* Renal failure (serum creatinine >200umol)
* Liver disease (ALT or AST >100 IU), especially acute hepatitis
* Hyperbilirubinemia
* Alcohol abuse
* Oral Anticoagulation
* Concomitant therapy with Phenobarbital, Phenytoin, Carbamazepin, Isonicotinic Acid, Chloramphenicol Chlorzoxazone, Zidovudine, Salicylamide
* Insulin-dependent diabetes mellitus
* Drug abuse
* Anemia (Hb<10 g/dl)
* Known allergies on Paracetamol
* Pregnancy
* Malignancy (unless healed or remission > 5 years)
* Symptomatic hypotension, hypertension >160/100 mmHg
* Disease with systemic inflammation (e.g. rheumatoid arthritis, M. Crohn)
* Participation in another study within the last month

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy endpoint: To investigate the effect of paracetamol on endothelial function as compared to placebo in patients with stable coronary artery disease. | 2 weeks
primary safety endpoint: to evaluate the effect of paracetamol on 24-hour systolic and diastolic blood pressure as compared to placebo in patients with stable coronary artery disease. | 2 Weeks

SECONDARY OUTCOMES:
To investigate the effect of paracetamol on markers of inflammation and oxidative stress as well as platelet function | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ruschitzka, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital, Zurich, Switzerland

REFERENCES:
- [Derived] Sudano I, Flammer AJ, Periat D, Enseleit F, Hermann M, Wolfrum M, Hirt A, Kaiser P, Hurlimann D, Neidhart M, Gay S, Holzmeister J, Nussberger J, Mocharla P, Landmesser U, Haile SR, Corti R, Vanhoutte PM, Luscher TF, Noll G, Ruschitzka F. Acetaminophen increases blood pressure in patients with coronary artery disease. Circulation. 2010 Nov 2;122(18):1789-96. doi: 10.1161/CIRCULATIONAHA.110.956490. Epub 2010 Oct 18. PMID 20956208